CLINICAL TRIAL: NCT06401980
Title: Addition of Darolutamide to First Line Treatment of Metastatic Castration-Resistant Prostate Cancer (mCRPC): a Randomized Open Label Phase II Trial
Brief Title: Darolutamide in Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 08/23
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; mCRPC; Darolutamide; phase II trial
MeSH Terms: interventions — darolutamide; Standard of Care

STUDY DESIGN:
Intervention Model Description: International, randomized, open label, phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Experimental (Experimental): Standard of Care
  + Darolutamide 2 x 600 mg BID until radiographic PD
  Interventions: Drug: Darolutamide
- Arm B: Control (Other): Standard of Care
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Darolutamide — Darolutamide will be supplied in bottles as 300 mg film-coated tablets for oral intake
  Other Names: Nubeqa®
  Arms: Arm A: Experimental
Other: Standard of care — * Docetaxel
  * Cabazitaxel
  * LuPSMA
  * Radium 223
  * Olaparib, in case of BRCA1 or 2 mutated or HRR deficient tumors
  The standard of care is chosen by the local investigator and respecting the country specific approvals.
  Arms: Arm B: Control

SUMMARY:
Despite improvements in treatment, metastatic prostate cancer remains incurable, especially in the case of pretreated metastatic castration-resistant disease (mCRPC), where treatment options are limited, leading to an unmet need. The paradigm shift in the treatment of metastatic hormone-sensitive prostate cancer (mHSPC) has affected the treatment landscape for mCRPC patients. Many have already received androgen deprivation therapy (ADT) and androgen receptor pathway inhibitors (ARPI), making first-line mCRPC treatment challenging.

The Swiss Group for Clinical Cancer Research (SAKK) has shown in previous studies that maintenance treatment with an ARPI, such as darolutamide, can improve radiographic progression-free survival (rPFS) in pretreated mCRPC patients. In the SAKK 08/16 trial, darolutamide maintenance was found to prolong PFS compared to placebo, especially in patients who responded well to prior ARPI treatment.

Based on these findings, the hypothesis is that continued AR-pathway blockade with darolutamide, initiated in patients progressing from mHSPC to mCRPC on ARPI treatment, can improve outcomes when added to standard first-line mCRPC therapy and continued as maintenance. The proposed study aims to evaluate the efficacy of darolutamide, combined with physician-choice standard of care (including taxane chemotherapy, olaparib, radium 223, or LuPSMA), followed by maintenance therapy, on rPFS for patients in the first-line setting of mCRPC.

DETAILED DESCRIPTION:
Metastatic prostate cancer remains incurable despite several major improvements in the treatment. In the case of pretreated metastatic castration-resistant disease (mCRPC) the options remain scarce and there is still an unmet need in this patient population.

For the majority of patients with metastatic hormone-sensitive prostate cancer (mHSPC) the combination of androgen deprivation (ADT) and ARPI (or even a triplet treatment with ADT, docetaxel and darolutamide or abiraterone) has become standard of care. However, when patients become metastatic castration resistant (mCRPC) over time a change of systemic treatment is necessary and thus this paradigm switch in treatment of mHSPC has had a major impact on treatment of mCRPC patients. Many patients developing metastatic castration-resistant disease these days have not only received ADT but also an ARPI and, in some cases, also docetaxel. Therefore, the treatment options in the first line setting of mCRPC are restricted and the outcome is poorer compared to the past. Improvement of first line mCRPC is an important unmet clinical need.

The SAKK has demonstrated in two earlier studies that maintenance treatment with an ARPI (orteronel in SAKK 08/11 or darolutamide in SAKK 08/16) can improve radiographic progression-free survival in pretreated mCRPC patients after ARPI and/or taxane based. This maintenance concept could be introduced more generally in the first line setting of mCRPC.

In the SAKK 08/16 trial, darolutamide maintenance was shown to prolong progression-free survival (PFS) compared to placebo, in patients with mCRPC who had received prior ARPI, and whose disease did not progress during taxane therapy. This benefit was more pronounced in patients with prior response to ARPI.

Taken together it is hypothesized that the continued AR-pathway blockade with darolutamide in patients progressing from mHSPC to mCRPC on ARPI treatment can improve outcome when it is added to a standard first line mCRPC therapy and then continued as maintenance. SAKK proposes to add the ARPI darolutamide to standard first line mCRPC treatment consisting of either taxane chemotherapy (docetaxel or cabazitaxel), olaparib, radium 223 or LuPSMA. The choice of standard of care treatment is up to the investigator, respecting the country specific approvals. Darolutamide will be given concomitantly with the chosen first line treatment and will be continued as maintenance afterwards until radiographic progression.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to Swiss law and ICH GCP E6(R2) regulations before registration and prior to any trial specific procedures
* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
* Castration resistance: tumor progression after orchiectomy or during treatment with GnRH analogues (agonists or antagonists).
* Non-surgically castrated patient agrees on ongoing use of GnRH analogues (agonists or antagonists) during the trial
* Metastatic disease, documented by imaging according to PCWG3 criteria
* Measurable disease or bone lesions that are evaluable according to PCWG3 criteria
* A minimum of 12 months on ADT+ARPI therapy (calculated from ADT initiation) within mHSPC setting, showing an at least 50% PSA response or partial remission according to RECIST v1.1. ARPI change within mHSPC is only allowed for intolerance.
* Progressive disease according to modified PCWG3 before registration is defined as (at least 2 out of 3):

  * PSA progression ≥ 25% above nadir (2 consecutive rises at least 3 weeks apart)
  * New metastatic lesion on imaging (at least two or more new bone lesions on bone scan or one new non-bone lesion or progression on PSMA-PET/CT according to PROMISE V2 criteria
  * Clinical progression
* Patients with a previously treated malignancy are eligible, when the risk of the prior malignancy interfering with either safety or efficacy endpoints is very low
* Age ≥ 18 years
* WHO performance status 0-2
* Adequate bone marrow function: absolute neutrophil count ≥ 1.0 x 109/L, platelet count ≥ 100 x 109/L, hemoglobin ≥ 90 g/L.
* Adequate hepatic function: total bilirubin ≤ 1.5 x ULN (except for patients with Gilbert's disease ≤ 3.0 x ULN), ALT and AST ≤ 2.5 x ULN, or ≤ 5 x ULN under the assumption that abnormal values are a result of cancer
* Adequate renal function: estimated glomerular filtration rate (eGFR) > 30 mL/min/1.73 m2 (according to CKD-EPI formula)
* Men agree not to donate sperm or to father a child during trial treatment and until 3 months after the last dose of trial treatment
* Patients are able and willing to swallow darolutamide as whole tablet.

Exclusion Criteria:

* Presence of a small cell component
* Prior systemic therapy for metastatic castration-resistant disease
* Prior chemotherapy for mHSPC, except docetaxel
* Prior LuPSMA or radium 223 for prostate cancer
* Concomitant or recent (within 28 days of registration) treatment with any other experimental drug
* Concomitant use of other anti-cancer drugs or radiotherapy except for local pain control and GnRH analogues
* Severe or uncontrolled cardiovascular disease
* Acute exacerbations of chronic illnesses, serious infections, or major surgery within 28 days before expected start of treatment
* Clinical or radiological evidence of current spinal cord compression
* Any concomitant drugs contraindicated for use with darolutamide according to the approved product information
* Known hypersensitivity to darolutamide
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the GI absorption or tolerance of darolutamide
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Radiographic progression-free survival (rPFS) | From the date of randomization until the date of radiographic disease progression or death from any cause, assessed up to 2 years after end of treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization until the date of death from any cause, assessed up to 2 years after end of treatment.
  OS is defined as the time from randomization until death due to any cause. Patients not experiencing an event (death) will be censored at the last date they were known to be alive.
Time to symptomatic/clinical progression | From date of randomization until the date of symptomatic/clinical progression, assessed up to 2 years after end of treatment
  Time to symptomatic/clinical progression is defined as the time from randomization to the time point of symptomatic/clinical progression. Patients not experiencing an event will be censored at the date of the last visit before initiation of a new anti-cancer treatment, if any.
  Symptomatic/clinical progression is defined by one of the following:
  * Occurrence of a SRE due to bone metastases, defined as pathologic fracture, spinal cord compression, palliative radiation to bone, or surgery to bone
  * Treating physician decides for intervention due to new disease related complications (e.g., urinary obstruction, hydronephrosis)
Time to PSA progression | From date of randomization until the date of PSA progression, assessed up to 2 years after end of treatment.
  Time to PSA progression is defined as the time from randomization to the time point of PSA progression. Patients not experiencing an event will be censored at the date of the last available PSA assessment before initiation of a new anti-cancer treatment, if any. PSA progression is defined as:
Event-free survival (EFS) | From date of randomization until the date of the event of interest, assessed up to 2 years after end of treatment.
  Event-free survival is defined as the time from randomization until the event of interest. Patients not experiencing an event will be censored at the date of the last available assessment before initiation of a new anti-cancer treatment, if any
Objective response rate according to RECIST | From the date of randomization until date of the end of treatment, estimated up to 2 years after registration
  Objective response is defined as any complete response (CR) or partial response (PR) according to RECIST 1.1 criteria (Appendix 1) achieved during treatment. Any patient with CR or PR as best observed response during treatment will be considered as a success; otherwise they will be considered as a failure.
  Patients without any tumor assessment or with non-evaluable response (NE) during treatment will be considered as failures for this endpoint.
PSA response (30%, 50%, 90% and best) | From the date of randomization until the end of treatment, estimated up to 2 years after registration.
Duration of PSA response (50%) | From the date of randomization until the date of PSA progression, assessed up to 2 years after end of treatment.
  Duration of PSA response is defined as the time from appearance of 50% PSA response during treatment to the time point of PSA progression. Definition of PSA progression is provided above. In case the patient does not experience PSA progression, the patient will be censored at the last PSA assessment before starting a new anti-cancer treatment, if any.
  This endpoint will be calculated for the subgroup of patients achieving 50% PSA response.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cathomas, Prof, Study Chair — Kantonsspital Graubünden; Ursula Vogl, MD, Study Chair — Istituto Oncologico della Svizzera Italiana
Locations (13):
- Switzerland (13):
  - Tumorzentrum Aarau TZA, Aarau
  - Kantonsspital Baden, Baden
  - Istituto Oncologico della Svizzera Italiana (IOSI), Bellinzona
  - Inselspital, Bern
  - Kantonsspital Graubuenden, Chur
  - Hôpitaux Universitaires Genève HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - OnkoZentrum Zürich - Standort Seefeld, Zurich
  - Stadtspital Triemli Zürich, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No